CLINICAL TRIAL: NCT02336711
Title: Molecular Imaging-based Dose Escalation in HPV Negative Patients With Locally Advanced Squamous Cell Carcinoma of the Oropharynx: a Phase-I Study.
Brief Title: Molecular Imaging-based Dose Escalation in HPV Negative Patients With Locally Advanced SCC of the Oropharynx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/13MAR/117
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation (Experimental): Dose escalation
  Interventions: Radiation: dose escalation

INTERVENTIONS:
Radiation: dose escalation — molecular imaging based radiotherapy dose escalation

SUMMARY:
Phase I study to assess the feasibility (i.e. early toxicity) of Molecular Imaging-based Dose Escalation in HPV Negative Patients With Locally Advanced SCC of the Oropharynx.

DETAILED DESCRIPTION:
The objective is to assess the feasibility (i.e. early toxicity) of an adaptive dose escalation through 18F-FDG-PET-based dose painting by numbers in 10 HPV negative patients with locally advanced squamous cell carcinoma of the oropharynx. Treatment will be delivered with Helical Tomotherapy® or volumetric-modulated arc therapy (VMAT). Dose adaptation will be performed at 2 time-points with per-treatment 18F-FDG-PET/CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with squamous cell carcinoma of the oropharynx, HPV-negative (p16 assay)
* T size of 3 cm or more in greatest dimension with the exclusion of tumor with bone infiltration
* N0, N1, N2a, N2b node (AJCC/UICC 7th edition)
* No distant metastasis
* No contra-indication to concomitant chemotherapy
* World Health Organization (WHO) Performance Status of 0 or 1 or Karnofsky performance status ≥ 80.
* Provision of written informed consent

Exclusion Criteria:

* Patients with induction chemotherapy will not be eligible
* Previous or concurrent history of cancer, except basal cell skin carcinoma
* Second primary tumor at the time of diagnosis
* Previous treatment with surgery, radiotherapy or chemotherapy for head and neck malignancy
* Any evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease), or psychological disorder
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | up to 3 months following the completion of radiotherapy

SECONDARY OUTCOMES:
Primary tumor control probability | at 1 and 2 years
Late toxicity | at 1 and 2 years
Progression-free survival | at 1 and 2 years
Overall survival | at 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Grégoire, MD, PhD, Principal Investigator — Department of Radiation Oncology, and Center for Molecular Imaging, Radiotherapy and Oncology (MIRO), Institut de Recherche Expérimentale et Clinique (IREC), Université catholique de Louvain, St-Luc University Hospital, Brussels, Belgium
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven